CLINICAL TRIAL: NCT02742974
Title: Fluid Resuscitation Optimization in Surgical Trauma Patients (FROST)
Acronym: FROST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-159
Record Dates: First submitted 2016-02-10; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Critical Illness; Trauma
Keywords: Trauma; Minimally Invasive Hemodynamic Monitoring; Perioperative; Complications; Hemodynamics; Operative procedures
MeSH Terms: conditions — Critical Illness; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FloTrac™ and EV1000™ pre and post-operatively (No Intervention): Cardiovascular management guided by minimally invasive hemodynamic monitoring via FloTrac™ and EV1000™ will be utilized in the pre and post-operative period in the control arm.
- FloTrac™ and EV1000™ peri-operatively (Experimental): Cardiovascular management guided by minimally invasive hemodynamic monitoring via FloTrac™ and EV1000™ will be utilized in the perioperative period for the intervention arm
  Interventions: Device: FloTrac™ and EV1000™

INTERVENTIONS:
Device: FloTrac™ and EV1000™ — Interventions to improve cardiovascular performance will be made in all patients whose cardiovascular function is sub-optimal in accordance with routine clinical management during trauma resuscitation. Patients who meet inclusion criteria will be assigned to the intervention or control arm of the study based on the process outlined in the protocol. Patients assigned to the intervention arm will have intra-operative hemodynamic monitoring performed by the anesthesia staff and cardiovascular interventions will be based off of the algorithm described in the protocol. Members of anesthesia or the surgical team can initiate interventions as indicated during routine ICU care or intra-operatively.
  Arms: FloTrac™ and EV1000™ peri-operatively

SUMMARY:
The aim of this study is to determine if the incidence of post-operative complications can be decreased by the implementation of intra-operative, minimally invasive hemodynamic monitoring (MIHM) via FloTrac™ and EV1000™ in trauma patients.

DETAILED DESCRIPTION:
Numerous factors are known to contribute to post-traumatic morbidity and mortality. Acute blood loss, hypovolemia, and systemic inflammatory response syndrome can often develop following severe traumatic injury and are, frequently, further exacerbated by the presence of pre-existing health conditions. The culmination of these insults and/or pre-existing conditions can precipitate an imbalance in oxygen delivery and consumption leading to tissue ischemia and resultant organ dysfunction.

Tissue ischemia precipitates a disruption in the balance of oxygen delivery and consumption often yielding a conversion from aerobic to anaerobic processes in order to maintain metabolic functionality. The conversion to anaerobic processes leads to the production of lactic acid and a resulting consumption of the body's basic buffers. Clinically, the consumption of the body's basic buffers is frequently referred to as the development of a base deficit. Both the production of lactic acid and the development of a base deficit have been positively linked to the increased morbidity and mortality in multiple critically ill patient populations, including those with traumatic injuries.

Multiple studies have linked the rate at which base deficit corrects or lactic acid clears to the likelihood of survival. Accordingly, hemodynamic monitoring can provide vital information concerning cardiovascular function including vascular volume, vascular capacitance, and cardiac performance. Obtaining this information enables clinicians to tailor interventions to target specific components of the cardiovascular system in order to most effectively reverse the cause of tissue hypoxia, elevation in lactic acid, and base deficit, while simultaneously decreasing the likelihood of causing harm through unnecessary or unwarranted changes in management.

Advancements in hemodynamic monitoring technology now allow clinicians to obtain data by using minimally invasive techniques. Devices utilizing this technology can be connected to vascular access routinely utilized in the intensive care setting such as arterial lines. These devices provide parameters such as systolic pressure variation (SPV), pulse pressure variation (PPV) and stroke volume variation (SVV) to predict fluid responsiveness of critically ill, mechanically ventilated patients. Studies evaluating these parameters have shown them to have a 84-94% positive predictive value for fluid responsiveness. In addition, higher variability in studied parameters were indicative of patients who were more likely to be responsive to fluid challenges.

Modern clinical management in critically ill patients with cardiovascular dysfunction hinges on reversal of the underlying cause of cardiovascular dysfunction. Recent management strategies have used a multi-faceted approach in which multiple processes of potential dysfunction can be monitored and managed simultaneously. Management is goal directed with clearly defined endpoints for the management of vascular volume, cardiac performance as well as maintenance of vascular capacitance. Hemodynamic monitoring technology is essential in providing data that will allow clinical interventions to be tailored to patient-specific physiology and provide goals for titration of therapy.

In recent years, data has emerged using goal directed therapy in the surgical patient population with favorable outcomes suggesting a decrease in post-operative organ dysfunction, ICU and hospital length of stay, however, there is limited data in the trauma patient population. This study endeavors to determine if the implementation of intra-operative monitoring will decrease the incidence of post-operative complications such as acute lung injury, infections, thromboembolism, cerebral vascular accident, acute kidney injury, myocardial infarction; in addition to the traditional outcome measures of mortality and length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Injury Severity Score > 15 (indicator of anticipated trauma mortality)
3. Admission to Surgical-Trauma ICU (STICU)
4. Anticipated surgery within 72 hours of admission
5. American Society of Anesthesiology patient classification status (ASA) 2-5
6. Lactic acid > 2.5 within 24 hours of surgical procedure or Base deficit ≥ - 5 mmol/L, or persistent requirement for vasopressor support within 24 hours of surgical procedure
7. Patient requires mechanical ventilation prior to consenting surgery
8. Vascular devices that include a minimum of an arterial line
9. Minimally invasive hemodynamic monitoring initiated prior to first surgical procedure unless patient is taken emergently, e.g. OR from trauma bay
10. Patients requiring emergent initial operative procedures will be eligible for consenting if above criteria are met prior to their second surgical procedure
11. Anticipated operative procedure precipitating evaluation and/or consenting for study must be > 30 minutes in duration

    * Procedures < 30 minutes would not result in significant metabolic stress necessitating a continuation of MIHM

Exclusion Criteria:

1. Pregnancy
2. Exclusions due to limitations with respect to accuracy of MIHM:

   * Patients not intubated prior to surgical procedure
   * Patients requiring an open thoracotomy
   * Patients with known history of surgical intervention for peripheral vascular disease
   * Patients with pre-existing atrial arrhythmias
   * Patients who are on cardiopulmonary bypass
3. Isolated acute cerebral injury and/or traumatic cerebral injury

   * Hemodynamic management in this patient population does not always follow typical/standard endpoints due to nuances of managing intracranial pressures
4. Cardiac arrest prior to enrollment
5. Patients with pre-existing, dialysis dependent, renal failure upon admission

   * Hemodynamic management in this patient population does not always follow typical/standard endpoints due to nuances of managing renal failure
6. Patients with pre-existing cirrhosis

   * Hepatic failure results in abnormal clearance of lactic acid
7. Patients with no survival injuries, e.g. gunshot wound to the head

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Complications | Post-operative complications during patient hospital stay up to 6 months
  The aim of this study is to determine if the incidence of post-operative complications will decreased with the implementation of intra-operative, minimally invasive hemodynamic monitoring via FloTrac™ and EV1000™ in trauma patients.

SECONDARY OUTCOMES:
Impact of Intervention | During patient hospital stay up to 6 months
  To evaluate the impact of continuing intra-operative minimally invasive hemodynamic monitoring via FloTrac™ and EV1000™ :
  * Intensive Care Unit (ICU) and hospital length of stay in days
  * Duration of post-operative vasopressor requirements in days
Impact of Intervention | During patient hospital stay up to 6 months
  To evaluate the impact of continuing intra-operative minimally invasive hemodynamic monitoring via FloTrac™ and EV1000™ :
  -ICU and hospital mortality rate
Lactic acid and Base deficit changes | Within 24 hours pre and post-surgery
  To compare the change in lactic acid and base deficit from the pre to post-operative period (most recent value within 24 hours pre and post-surgery). Both lactic acid and base deficit values will be recorded in mmoL/L.
APACHE II | Within 24 hours pre and post-surgery
  Acute Physiology and Chronic Health Evaluation (APACHE) II score between study cohorts. These scores will be recorded in whole numbers.
SOFA scores | Within 24 hours pre and post-surgery
  Sepsis-related Organ Failure (SOFA) score between study cohorts. These scores will be recorded in whole numbers.
Changes in pre and post-operative lactic acid and base deficit | Within 24 hours pre and post-surgery
  To compare changes in pre and post-operative lactic acid and based deficit between cohorts based on duration of surgical interventions. Both lactic acid and base deficit values will be recorded in mmoL/L.
Changes in pre and post-operative APACHE II score | Within 24 hours pre and post-surgery
  To compare changes in pre and post-operative APACHE II scores between cohorts based on duration of surgical interventions. This score will be recorded in whole numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Audis Bethea, PharmD, BCPS, Principal Investigator — CAMC Health System
Locations (1):
- Charleston Area Medical Center, General Hospital, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Husain FA, Martin MJ, Mullenix PS, Steele SR, Elliott DC. Serum lactate and base deficit as predictors of mortality and morbidity. Am J Surg. 2003 May;185(5):485-91. doi: 10.1016/s0002-9610(03)00044-8. PMID 12727572
- [Result] Abramson D, Scalea TM, Hitchcock R, Trooskin SZ, Henry SM, Greenspan J. Lactate clearance and survival following injury. J Trauma. 1993 Oct;35(4):584-8; discussion 588-9. doi: 10.1097/00005373-199310000-00014. PMID 8411283
- [Result] Cerovic O, Golubovic V, Spec-Marn A, Kremzar B, Vidmar G. Relationship between injury severity and lactate levels in severely injured patients. Intensive Care Med. 2003 Aug;29(8):1300-5. doi: 10.1007/s00134-003-1753-8. Epub 2003 Jul 9. PMID 12904861
- [Result] Arnold RC, Shapiro NI, Jones AE, Schorr C, Pope J, Casner E, Parrillo JE, Dellinger RP, Trzeciak S; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Multicenter study of early lactate clearance as a determinant of survival in patients with presumed sepsis. Shock. 2009 Jul;32(1):35-9. doi: 10.1097/shk.0b013e3181971d47. PMID 19533847
- [Result] Nguyen HB, Rivers EP, Knoblich BP, Jacobsen G, Muzzin A, Ressler JA, Tomlanovich MC. Early lactate clearance is associated with improved outcome in severe sepsis and septic shock. Crit Care Med. 2004 Aug;32(8):1637-42. doi: 10.1097/01.ccm.0000132904.35713.a7. PMID 15286537
- [Result] Callaway DW, Shapiro NI, Donnino MW, Baker C, Rosen CL. Serum lactate and base deficit as predictors of mortality in normotensive elderly blunt trauma patients. J Trauma. 2009 Apr;66(4):1040-4. doi: 10.1097/TA.0b013e3181895e9e. PMID 19359912
- [Result] Dunne JR, Tracy JK, Scalea TM, Napolitano LM. Lactate and base deficit in trauma: does alcohol or drug use impair their predictive accuracy? J Trauma. 2005 May;58(5):959-66. doi: 10.1097/01.ta.0000158508.84009.49. PMID 15920409
- [Result] Ouellet JF, Roberts DJ, Tiruta C, Kirkpatrick AW, Mercado M, Trottier V, Dixon E, Feliciano DV, Ball CG. Admission base deficit and lactate levels in Canadian patients with blunt trauma: are they useful markers of mortality? J Trauma Acute Care Surg. 2012 Jun;72(6):1532-5. doi: 10.1097/TA.0b013e318256dd5a. PMID 22695417
- [Result] Ziegler DW, Wright JG, Choban PS, Flancbaum L. A prospective randomized trial of preoperative "optimization" of cardiac function in patients undergoing elective peripheral vascular surgery. Surgery. 1997 Sep;122(3):584-92. doi: 10.1016/s0039-6060(97)90132-x. PMID 9308617
- [Result] Landry DW, Oliver JA. The pathogenesis of vasodilatory shock. N Engl J Med. 2001 Aug 23;345(8):588-95. doi: 10.1056/NEJMra002709. No abstract available. PMID 11529214
- [Result] Otero RM, Nguyen HB, Huang DT, Gaieski DF, Goyal M, Gunnerson KJ, Trzeciak S, Sherwin R, Holthaus CV, Osborn T, Rivers EP. Early goal-directed therapy in severe sepsis and septic shock revisited: concepts, controversies, and contemporary findings. Chest. 2006 Nov;130(5):1579-95. doi: 10.1378/chest.130.5.1579. PMID 17099041
- [Result] Monnet X, Dres M, Ferre A, Le Teuff G, Jozwiak M, Bleibtreu A, Le Deley MC, Chemla D, Richard C, Teboul JL. Prediction of fluid responsiveness by a continuous non-invasive assessment of arterial pressure in critically ill patients: comparison with four other dynamic indices. Br J Anaesth. 2012 Sep;109(3):330-8. doi: 10.1093/bja/aes182. Epub 2012 Jun 26. PMID 22735299
- [Result] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Result] Vincent JL, Weil MH. Fluid challenge revisited. Crit Care Med. 2006 May;34(5):1333-7. doi: 10.1097/01.CCM.0000214677.76535.A5. PMID 16557164
- [Result] Osman D, Ridel C, Ray P, Monnet X, Anguel N, Richard C, Teboul JL. Cardiac filling pressures are not appropriate to predict hemodynamic response to volume challenge. Crit Care Med. 2007 Jan;35(1):64-8. doi: 10.1097/01.CCM.0000249851.94101.4F. PMID 17080001
- [Result] Mythen MG, Webb AR. Perioperative plasma volume expansion reduces the incidence of gut mucosal hypoperfusion during cardiac surgery. Arch Surg. 1995 Apr;130(4):423-9. doi: 10.1001/archsurg.1995.01430040085019. PMID 7535996
- [Result] Bishop MH, Shoemaker WC, Appel PL, Meade P, Ordog GJ, Wasserberger J, Wo CJ, Rimle DA, Kram HB, Umali R, et al. Prospective, randomized trial of survivor values of cardiac index, oxygen delivery, and oxygen consumption as resuscitation endpoints in severe trauma. J Trauma. 1995 May;38(5):780-7. doi: 10.1097/00005373-199505000-00018. PMID 7760409
- [Result] Buettner M, Schummer W, Huettemann E, Schenke S, van Hout N, Sakka SG. Influence of systolic-pressure-variation-guided intraoperative fluid management on organ function and oxygen transport. Br J Anaesth. 2008 Aug;101(2):194-9. doi: 10.1093/bja/aen126. Epub 2008 May 28. PMID 18511439
- [Result] Benes J, Chytra I, Altmann P, Hluchy M, Kasal E, Svitak R, Pradl R, Stepan M. Intraoperative fluid optimization using stroke volume variation in high risk surgical patients: results of prospective randomized study. Crit Care. 2010;14(3):R118. doi: 10.1186/cc9070. Epub 2010 Jun 16. PMID 20553586
- [Result] Lobo SM, Lobo FR, Polachini CA, Patini DS, Yamamoto AE, de Oliveira NE, Serrano P, Sanches HS, Spegiorin MA, Queiroz MM, Christiano AC Jr, Savieiro EF, Alvarez PA, Teixeira SP, Cunrath GS. Prospective, randomized trial comparing fluids and dobutamine optimization of oxygen delivery in high-risk surgical patients [ISRCTN42445141]. Crit Care. 2006;10(3):R72. doi: 10.1186/cc4913. Epub 2006 May 12. PMID 16696864
- [Result] Chytra I, Pradl R, Bosman R, Pelnar P, Kasal E, Zidkova A. Esophageal Doppler-guided fluid management decreases blood lactate levels in multiple-trauma patients: a randomized controlled trial. Crit Care. 2007;11(1):R24. doi: 10.1186/cc5703. PMID 17313691
- [Result] McKendry M, McGloin H, Saberi D, Caudwell L, Brady AR, Singer M. Randomised controlled trial assessing the impact of a nurse delivered, flow monitored protocol for optimisation of circulatory status after cardiac surgery. BMJ. 2004 Jul 31;329(7460):258. doi: 10.1136/bmj.38156.767118.7C. Epub 2004 Jul 8. PMID 15242867
- [Result] Lobo SM, Ronchi LS, Oliveira NE, Brandao PG, Froes A, Cunrath GS, Nishiyama KG, Netinho JG, Lobo FR. Restrictive strategy of intraoperative fluid maintenance during optimization of oxygen delivery decreases major complications after high-risk surgery. Crit Care. 2011;15(5):R226. doi: 10.1186/cc10466. Epub 2011 Sep 23. PMID 21943111
- [Result] Donati A, Loggi S, Preiser JC, Orsetti G, Munch C, Gabbanelli V, Pelaia P, Pietropaoli P. Goal-directed intraoperative therapy reduces morbidity and length of hospital stay in high-risk surgical patients. Chest. 2007 Dec;132(6):1817-24. doi: 10.1378/chest.07-0621. Epub 2007 Oct 9. PMID 17925428
- [Result] Arkilic CF, Taguchi A, Sharma N, Ratnaraj J, Sessler DI, Read TE, Fleshman JW, Kurz A. Supplemental perioperative fluid administration increases tissue oxygen pressure. Surgery. 2003 Jan;133(1):49-55. doi: 10.1067/msy.2003.80. PMID 12563237
- [Result] Polonen P, Ruokonen E, Hippelainen M, Poyhonen M, Takala J. A prospective, randomized study of goal-oriented hemodynamic therapy in cardiac surgical patients. Anesth Analg. 2000 May;90(5):1052-9. doi: 10.1097/00000539-200005000-00010. PMID 10781452
- [Result] Abbas SM, Hill AG. Systematic review of the literature for the use of oesophageal Doppler monitor for fluid replacement in major abdominal surgery. Anaesthesia. 2008 Jan;63(1):44-51. doi: 10.1111/j.1365-2044.2007.05233.x. PMID 18086070
- [Result] Wakeling HG, McFall MR, Jenkins CS, Woods WG, Miles WF, Barclay GR, Fleming SC. Intraoperative oesophageal Doppler guided fluid management shortens postoperative hospital stay after major bowel surgery. Br J Anaesth. 2005 Nov;95(5):634-42. doi: 10.1093/bja/aei223. Epub 2005 Sep 9. PMID 16155038
- [Result] Noblett SE, Snowden CP, Shenton BK, Horgan AF. Randomized clinical trial assessing the effect of Doppler-optimized fluid management on outcome after elective colorectal resection. Br J Surg. 2006 Sep;93(9):1069-76. doi: 10.1002/bjs.5454. PMID 16888706
- [Result] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Result] Venn R, Steele A, Richardson P, Poloniecki J, Grounds M, Newman P. Randomized controlled trial to investigate influence of the fluid challenge on duration of hospital stay and perioperative morbidity in patients with hip fractures. Br J Anaesth. 2002 Jan;88(1):65-71. doi: 10.1093/bja/88.1.65. PMID 11881887
- [Result] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Result] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Result] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- See also: SOFA Calculator — http://clincalc.com/IcuMortality/SOFA.aspx
- See also: APACHE II Calculator — http://clincalc.com/IcuMortality/APACHEII.aspx